CLINICAL TRIAL: NCT00320515
Title: Phase 1/2 Study of Pemetrexed Plus Cisplatin in Unresectable, Advanced Gastric Carcinoma.
Brief Title: Study of Pemetrexed Plus Cisplatin in Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7461; H3E-AA-S038
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-08

CONDITIONS: Neoplasm, Gastric
MeSH Terms: conditions — Stomach Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — Phase 1 - dose escalating: 600 mg/m2 level 1, 700 mg/m2 level 2, 800 mg/m2 level 3, 900 mg/m2 level 4, intravenous (IV), every 21 days, until disease progression
  Phase 2 - 700 mg/m2, intravenous (IV), every 21 days, until disease progression
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m2, intravenous (IV), every 21 days, until disease progression

SUMMARY:
This is a multicenter, single arm, open-label Phase 1/2 study of pemetrexed plus cisplatin for patients with unresectable, advanced gastric cancer who had no prior palliative chemotherapy. Phase 1 was designed to determine the optimal dose of pemetrexed for its phase 2, which has been completed and now a total of 60 qualified patients will be enrolled in the phase 2 of this study. The treating physician will determined the maximum number of cycles of pemetrexed plus cisplatin that a patient may receive in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven diagnosis of adenocarcinoma of the stomach
* Stage IV disease not amenable to curative surgery.
* Disease status must be that of measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate organ functions

Exclusion Criteria:

* Prior palliative chemotherapy for advanced gastric cancer.
* Pregnancy and breast feeding.
* Known or suspected brain metastasis and secondary primary malignancy
* Inability to interrupt aspirin, or other non-steroidal anti-inflammatory agents for a 5-day period.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.
* Concurrent administration of any other tumor therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559, Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucumain
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Obregón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a Phase 1/2 trial. There were 16 participants in Phase 1. None of them qualified for the Phase 2 portion of the trial. There were 73 participants in Phase 2; however, 4 were excluded from all analyses due to data quality issues at one site. Results presented here are for the 69 participants in Phase 2.
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 700 mg/m2, intravenous (IV), every 21 days, until disease progression Cisplatin: 75 mg/m2, intravenous (IV), every 21 days, until disease progression
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 69
Completed | 20
Not Completed | 49
Not completed — Death | 33
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 69
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 49
Region of Enrollment [Number; unit: participants]
  Taiwan | 22
  Mexico | 4
  Argentina | 18
  Korea, Republic of | 25
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 42
    1 - Ambulatory, Restricted Strenuous Activity | 27
Race/Ethnicity [Number; unit: participants]
  Caucasian | 1
  East Asian | 47
  Hispanic | 21

OUTCOME MEASURES:

1. Primary Outcome: Objective Best Tumor Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to measured progressive disease (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until disease progression, or up to 12 months after enrollment)
Population: All enrolled participants who received at least one dose of study drug. One participant was excluded from analysis because of no measurable disease at baseline.
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 68
participants
  Complete Response | 1
  Partial Response | 15
  Stable Disease | 22
  Progressive Disease | 24
  Unknown | 6

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of response to progressive disease or death (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until disease progression, or up to 12 months after enrollment)
Population: All enrolled participants who received at least one dose of study drug, had measureable disease at baseline, and had confirmed complete or partial responses. There were 16 patients qualified for the analysis of duration of response. Twelve participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 16
months | 5.4 [4.6 to 6.9]

3. Secondary Outcome: Progression Free Survival
Description: The period from study entry until disease progression or death on study, whichever occurred first.
Time Frame: baseline to measured progressive disease or death (Tumor assessments were performed every 2 cycles during therapy and 6-8 weeks during post-therapy until disease progression, or up to 12 months after enrollment)
Population: All enrolled participants who received at least one dose of study drug and had measureable disease at baseline. Twenty-six participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 68
months | 4.9 [2.8 to 7.1]

4. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact.
Time Frame: baseline to date of death from any cause (Survival follow-up were performed every 2 cycles during therapy and approximately every 3 months during post-therapy until death or up to 12 months after enrollment)
Population: All enrolled participants who received at least one dose of study drug and had measurable disease at baseline. Thirty-five participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 68
months | 11.8 [7.2 to 18.5]

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 14
Other Adverse Events (participants affected / at risk) | 69
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Neutropenia (Blood and lymphatic system disorders) | 1/69 (1)
Abdominal pain (Gastrointestinal disorders) | 1/69 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1/69 (1)
Ascites (Gastrointestinal disorders) | 1/69 (1)
Colonic obstruction (Gastrointestinal disorders) | 1/69 (1)
Ileus (Gastrointestinal disorders) | 2/69 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2/69 (2)
Vomiting (Gastrointestinal disorders) | 1/69 (1)
Dehydration (Metabolism and nutrition disorders) | 1/69 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/69 (1)
Central nervous system lesion (Nervous system disorders) | 1/69 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1/69 (1)
Renal failure (Renal and urinary disorders) | 1/69 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1/69 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/69 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/69 (1)
Deep vein thrombosis (Vascular disorders) | 1/69 (1)
Hypotension (Vascular disorders) | 1/69 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 13/69 (24)
Leukopenia (Blood and lymphatic system disorders) | 6/69 (9)
Lymphopenia (Blood and lymphatic system disorders) | 12/69 (18)
Neutropenia (Blood and lymphatic system disorders) | 22/69 (43)
Abdominal distension (Gastrointestinal disorders) | 8/69 (9)
Abdominal pain (Gastrointestinal disorders) | 13/69 (14)
Constipation (Gastrointestinal disorders) | 24/69 (32)
Diarrhoea (Gastrointestinal disorders) | 16/69 (24)
Dyspepsia (Gastrointestinal disorders) | 4/69 (4)
Nausea (Gastrointestinal disorders) | 37/69 (89)
Stomatitis (Gastrointestinal disorders) | 4/69 (7)
Vomiting (Gastrointestinal disorders) | 26/69 (51)
Asthenia (General disorders) | 6/69 (6)
Fatigue (General disorders) | 29/69 (52)
Mucosal inflammation (General disorders) | 4/69 (6)
Oedema (General disorders) | 5/69 (5)
Alanine aminotransferase increased (Investigations) | 6/69 (6)
Aspartate aminotransferase increased (Investigations) | 8/69 (9)
Blood alkaline phosphatase increased (Investigations) | 12/69 (17)
Blood bilirubin increased (Investigations) | 4/69 (4)
Blood creatinine increased (Investigations) | 7/69 (18)
Creatinine renal clearance decreased (Investigations) | 4/69 (4)
Haemoglobin decreased (Investigations) | 30/69 (45)
Neutrophil count decreased (Investigations) | 26/69 (65)
Platelet count decreased (Investigations) | 11/69 (21)
Weight decreased (Investigations) | 10/69 (11)
White blood cell count decreased (Investigations) | 18/69 (27)
Anorexia (Metabolism and nutrition disorders) | 27/69 (56)
Decreased appetite (Metabolism and nutrition disorders) | 6/69 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 4/69 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5/69 (12)
Hyperglycaemia (Metabolism and nutrition disorders) | 14/69 (30)
Hyperkalaemia (Metabolism and nutrition disorders) | 11/69 (14)
Hypocalcaemia (Metabolism and nutrition disorders) | 9/69 (19)
Hypokalaemia (Metabolism and nutrition disorders) | 4/69 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5/69 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 13/69 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 7/69 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 6/69 (8)
Dizziness (Nervous system disorders) | 10/69 (19)
Headache (Nervous system disorders) | 10/69 (14)
Hypoaesthesia (Nervous system disorders) | 7/69 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 6/69 (6)
Insomnia (Psychiatric disorders) | 9/69 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 11/69 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8/69 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 9/69 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4/69 (4)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 10/69 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7/69 (9)
Rash (Skin and subcutaneous tissue disorders) | 7/69 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days